CLINICAL TRIAL: NCT05707325
Title: A Multicenter, Single-arm, Open-label, Dose-escalation and Dose-expansion Clinical Study Evaluating the Safety, Tolerability and Preliminary Efficacy of Engineered Red Blood Cell in Patients With Advanced Malignancies
Brief Title: Safety, Tolerability and Preliminary Efficacy of Engineered Red Blood Cell in Patients With Advanced Malignancies
Acronym: Reboot-101
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Westlake Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Reboot-101
Record Dates: First submitted 2023-01-11; First posted 2023-01-31 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Cancer; Solid Tumor; Hematologic Malignancy
Keywords: solid tumors; hematologic malignancies
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: The dose escalation part is carried out according to the "3+3" increasing principle. At least four dose groups are predefined based on the number of engineered red blood cells, specifically 1e11, 2e11, 3e11, 3.5e11,etc.
  Dose expansion part will be decided according to dose escalation part.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose Escalation in Solid tumors and Hematologic malignancies (Experimental): In Dose Escalation part， all patients will be enrolled in different doses according to the Study Protocol for evaluate the recommend dose
  Interventions: Drug: engineered red blood cell
- Dose Expansion in Solid tumors and Hematologic malignancies (Experimental): In Expansion part， all patients will be enrolled in recommended dose
  Interventions: Drug: engineered red blood cell

INTERVENTIONS:
Drug: engineered red blood cell — engineered red blood cell

SUMMARY:
This is an investigator-initiated trial aimed at evaluating the safety and preliminary efficacy of a novel red blood cell-based therapy, where engineered red blood cells are conjugated with checkpoint inhibitors.

DETAILED DESCRIPTION:
The present study has 2 parts，including dose escalation and dose expansion。The dose escalation part is carried out according to the "3+3" increasing principle. At least four dose groups are predefined based on the number of engineered red blood cells, specifically 1e11, 2e11, 3e11, 3.5e11,etc.

Dose expansion part will be decided according to dose escalation part.

ELIGIBILITY:
Inclusion Criteria:

* 1.Histologically- or cytologically-proven advanced malignancies;
* 2.Male or female, 18 years of age or older but no more than 75 at the time of signing informed consent;
* 3.Dose escalation stage: (1) patients with advanced solid tumors who have received at least 2 regimens, and PDx monotherapy or combination therapy is included in the last regimen ; or patients received 1st regimen or above who cannot tolerate standard therapy but PDx monotherapy or combination therapy should be included in the last regimen.(2)Patients with relapsed and refractory malignant lymphomas (including: classic Hodgkin lymphoma (cHL), primary mediastinal large B-cell lymphoma PMBCL , Extranodal NK/T-cell lymphoma ENKTCL, mycosis fungoides/Sezari syndrome MF/SS) , or patients have no standard therapy, or are unable to receive standard therapy, PDx monotherapy or combination therapy is used in the last regimen.(3)All patients did not receive systemic therapy after disease progression and the time of disease progression cannot exceed 3 months, radiotherapy was acceptable (definition of secondary resistance: achieved disease control (including CR/PR/ SD), but then disease progression after PDx therapy);
* 4.Dose expansion stage:(1)patients with advanced solid tumors who have received at least 1 regimen or these is no standard systematic therapy or patients can not recieve standard therapy, but PDx monotherapy or combination therapy should be included in the last regimen.(2)patients with relapsed and refractory malignant lymphomas who have no standard therapy or can not receive standard therapy, but PDx monotherapy or combination therapy should be included in the last regimen.(3)All patients did not receive systemic therapy after disease progression and the time of disease progression cannot exceed 3 months, radiotherapy was acceptable (definition of secondary resistance: achieved disease control (including CR/PR/ SD), but then disease progression after PDx therapy);
* 5.Solid tumor：at least one lesion that is measurable according to RECIST 1.1;lymphomas:at least one visble or evaluable lesion that is measurable according to Lugano2014;
* 6.Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1;
* 7.Take the shorter one as the washout period before experimental treatment (28 days after the last tumor treatment, or 5 half lives);
* 8.Resolution of all acute reversible toxic effects of prior therapy or surgical procedure to baseline or Grade ≤1 (except alopecia and peripheral neurotoxicity);
* 9.Adequate organ function;
* 10.Estimated life expectancy of ≥12 weeks;
* 11.Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF).

Exclusion Criteria:

* 1.Any active or recently diagnosed clear or suspected autoimmune disorder disease;
* 2. Other serious medical diseases, including but not limited to: uncontrolled diabetes, active peptic ulcer, liver cirrhosis, active bleeding, etc., and those with uncontrolled or serious cardiovascular disease, such as the NYHA II or higher heart failure, unstable angina, myocardial infarction and other cardiovascular disease within 6 months before first administration, and uncontrolled hypertension (systolic blood pressure ≥ 180 mmHg and/or diastolic blood pressure ≥ 100 mmHg);
* 3.Has known active Hepatitis B or Hepatitis C or HIV;
* 4.Active brain metastases and/or cancerous meningitis;
* 5.Known history of any diseases affecting the quality and stability of erythropoiesis;
* 6.The spleen has been removed or, as judged by the investigator, a splenectomy may be planned during the trial;
* 7.Received at least one alive virus vaccination within 6 months before the first dose (except for the COVID-19 inactivated vaccine);
* 8.Known history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, severely impaired lung function, etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Dose-Limiting Toxicities (DLTs) According to National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI-CTCAE v.5.0) in Participants in escalating part. | 21 days
  DLTs were assessed according to NCI-CTCAE v.5.0 during the first cycle (21 days) and were defined as occurrence of any of the following toxicities if judged by the investigator to be possibly, probably or definitely related to study drug administration。
Number of Participants Who Experienced an Adverse Event (AE) | Up to approximately 24 months
  An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the Sponsor's product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition which was temporally associated with the use of the Sponsor's product was also an AE. The number of participants who experienced an AE was reported for all patients.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) According to Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1) | per 6 weeks
  ORR was defined as the percentage of participants in the analysis population who had a confirmed Complete Response (CR: disappearance of all lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters [SOD] of target lesions, taking as reference the baseline SOD) according to RECIST 1.1(only for solid tumor) or Lugano2014( only for lymphomas)
Anti-drug antibody (ADA) | 1 year
  Describe the number and percentage of anti-drug antibodies (ADA) produced by subjects at each time point after treatment, and the time of producing ADA.
Maximum Concentration (Cmax) of engineered red blood cells in all Participants | Cycle 1: Pre-dose, post-dose at 0.5, 6 and 12 hours and Days 2, 3, 8 and 15
  Blood samples were collected at specified intervals for the determination of Cmax. Cmax was defined as the maximum concentration of engineered red blood cells reached. Cmax was based on noncompartmental analysis and reported for all participants
Time to Maximum Concentration (Tmax) f engineered red blood cells in all Participants | Cycle 1: Pre-dose, post-dose at 0.5, 6 and 12 hours and Days 2, 3, 8 and 15
  Blood samples were collected at specified intervals for the determination of Tmax. Tmax was defined as time to the maximum concentration of engineered red blood cells reached. Tmax was based on noncompartmental analysis and reported for all participants

CONTACTS AND LOCATIONS:
Overall Officials: xiangmin Tong, Phd, Principal Investigator — ZHEJIANG PROVINCIAL PEOPLE'S HOSPITAL of China
Locations (1):
- Zhejiang Provincial People'S Hospital, Hangzhou, Zhejiang, China